CLINICAL TRIAL: NCT03558724
Title: Fluorescence Molecular Endoscopy of Locally Advanced Esophageal Carcinoma Using Bevacizumab-800CW to Evaluate Dose Response After Neoadjuvant Chemoradiotherapy: a Single-center Feasibility Study.
Brief Title: Fluorescence Endoscopy of Esophageal Carcinoma
Acronym: ORCA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose-escalation was finished, but no clear correlation between fluorescence and tumor grade was established
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL65856.042.18
Record Dates: First submitted 2018-05-17; First posted 2018-06-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer
Keywords: Fluorescence; Endoscopy; Bevacizumab-800CW; Locally advanced esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIR endoscopy with 4.5 mg bevacizumab-800CW (Experimental): A non-randomized, non-blinded, prospective, feasibility study.
  * IV-administration of 4.5 mg of the fluorescent tracer bevacizumab-800CW to a total of 5 patients with locally advanced esophageal cancer. The optimal dose will be expanded to include 30 patients.
  * Molecular fluorescence endoscopy: 2-3 days after administration, molecular fluorescence endoscopy will be performed with additional measurements of fluorescence signals.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform
- NIR endoscopy with 10 mg bevacizumab-800CW (Experimental): A non-randomized, non-blinded, prospective, feasibility study.
  * IV-administration of 10 mg of the fluorescent tracer bevacizumab-800CW to a total of 3 patients with locally advanced esophageal cancer. The optimal dose will be expanded to include 30 patients.
  * Molecular fluorescence endoscopy: 2-3 days after administration, molecular fluorescence endoscopy will be performed with additional measurements of fluorescence signals.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform
- NIR endoscopy with 25 mg bevacizumab-800CW (Experimental): A non-randomized, non-blinded, prospective, feasibility study.
  * IV-administration of 25 mg of the fluorescent tracer bevacizumab-800CW to a total of 3 patients with locally advanced esophageal cancer. The optimal dose will be expanded to include 30 patients.
  * Molecular fluorescence endoscopy: 2-3 days after administration, molecular fluorescence endoscopy will be performed with additional measurements of fluorescence signals.
  Interventions: Drug: Bevacizumab-IRDye800CW; Device: Molecular Fluorescence Endoscopy platform

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — Intravenous administration of 4.5, 10 or 25 mg of Bevacizumab-IRDye800CW prior to the endoscopic procedure
  Other Names: Tracer administration
Device: Molecular Fluorescence Endoscopy platform — A flexible fluorescence fiber-bundle is attached to a fluorescence camera platform to enable the detection of fluorescence signals. The fluorescence fiber-probe is inserted through the standard working channel of the standard clinical endoscope. Fluorescence imaging will be performed prior to and post the chemoradiotherapy.
  Other Names: Fluorescence Endoscopy

SUMMARY:
For locally advanced esophageal cancer (EC), neoadjuvant chemoradiotherapy (nCRT) for 5 weeks followed by esophagectomy and lymphadenectomy, if necessary, is standard of care. It is reported that the pathological complete response (pCR) rate after nCRT ranges from 16% to 43%, with a median of 26.5%. According to current clinical guidelines, patients who achieved pCR still go for surgery even though those patients who achieved pCR may not benefit from surgery. Besides, about 50% of EC patients may have post-operative complications including pneumonia, anastomotic leakage, recurrent laryngeal nerve paralysis, which lead to low health-related quality of life (HQoL).

The golden standard to test the pathological response is by pathological assessment of the surgical specimen and thus after surgery. Theoretically, if pCR after nCRT can be predicted accurately before surgery by advanced imaging techniques, patients could have a wait-and-see. The wait-and-see procedure includes regular follow-up and salvage surgery if recurrence is present. Therefore, molecular fluorescence endoscopy (FME) using near-infrared fluorescence (NIRF) tracer bevacizumab-800CW targeting vascular endothelial growth factor combined with high-definition white light (HD-WL) endoscopy is expected to be a promising technique to monitor pCR and fill the gap.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced esophageal carcinoma (cT1b-4a N0-3 M0) in multi-disciplinary esophageal oncology meeting agreed on long course neoadjuvant chemoradiotherapy, followed by esophagectomy;
* Age ≥ 18 years;
* Written informed consent.

Exclusion Criteria:

* Patients with psychological diseases or medical issues who are not able to sign informed consent form;

  * Concurrent uncontrolled medical conditions;
  * Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);
  * Irradical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of primary tumor prior to start of neoadjuvant chemoradiotherapy
  * Received a different investigational drug within 30 days prior to the dose of bevacizumab-800CW;
  * History of infusion reactions to bevacizumab or other monoclonal antibodies;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Discrimination of tumorous and non-tumorous tissue based on in vivo and ex vivo fluorescence measurements from bevacizumab-800CW gained during fluorescence endoscopy procedure | Three days after tracer injection
  To determine the sensitivity of the marker bevacizumab-800CW in discriminating between tumorous and non-tumorous tissue prior to and post neoadjuvant chemoradiotherapy, to identify patients who benefit from the chemoradiotherapy.
Safety of bevacizumab-800CW administration by monitoring vital signs and/or (serious) adverse events. | Up to 14 days after tracer injection
  Monitoring vital signs (blood pressure, heart frequency and temperature) and/or (serious) adverse events that are related to the administration of bevacizumab-800CW

SECONDARY OUTCOMES:
The correlation of in vivo and ex vivo fluorescent signals to histopathological analysis results | Up to 1,5 year
  Correlate the H/E images to the fluorescent images made with multiple ex vivo imaging modalities.
Quantification of the fluorescent signal by MDSFR/SFF spectroscopy | Up to 1,5 year
  Multi-diameter single-fiber reflectance with single-fiber fluorescence (MDSFR/SFF) spectroscopy can measure the fluorescence signal quantitatively, both in vivo and ex vivo.
To localization and distribution of bevacizumab-800CW fluorescent signal at cell level observed in vivo by confocal laser endomicroscopy (CLE) | Up to 1,5 year
  CLE is a confocal laser endomicroscopy system which enables in vivo microscopic images of the tissue
Assessment of the (sub)-cellular distribution of bevacizumab-800CW by ex vivo fluorescence microscopy | Up to 1,5 year
  Imaging of the distribution of bevacizumab-800CW with a fluorescence microscoop.
The variation in fluorescence intensity between fluorescence molecular endoscopy before and after neoadjuvant chemoradiotherapy defined as the tumor to background ratio and intrinsic fluorescence. | Up to 1,5 year
  Both the images and specific measurements are used to calculate the fluorescence intensity (TBR & intrinsic fluorescence) and a difference between the before and after intensity is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: W. B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen; G. M. van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duan XF, Tang P, Yu ZT. Neoadjuvant chemoradiotherapy for resectable esophageal cancer: an in-depth study of randomized controlled trials and literature review. Cancer Biol Med. 2014 Sep;11(3):191-201. doi: 10.7497/j.issn.2095-3941.2014.03.005. PMID 25364580
- [Background] Booka E, Takeuchi H, Nishi T, Matsuda S, Kaburagi T, Fukuda K, Nakamura R, Takahashi T, Wada N, Kawakubo H, Omori T, Kitagawa Y. The Impact of Postoperative Complications on Survivals After Esophagectomy for Esophageal Cancer. Medicine (Baltimore). 2015 Aug;94(33):e1369. doi: 10.1097/MD.0000000000001369. PMID 26287423
- [Background] Raymond D. Complications of esophagectomy. Surg Clin North Am. 2012 Oct;92(5):1299-313. doi: 10.1016/j.suc.2012.07.007. PMID 23026283